CLINICAL TRIAL: NCT07236684
Title: Identification of Factors Related to Urinary Incontinence in Patients With Multiple Sclerosis and Electromyographic Assessment of Pelvic Floor Muscle Activity: A Cross-Sectional Study
Brief Title: Identification of Factors Related to UI in Patients With MS and EMG Assessment of PFM Activity
Status: Not yet recruiting | Type: Observational
Sponsor: Artvin Coruh University (Other)
Responsible Party: Principal Investigator, Zeynep Yıldız Kızkın, Lecturer, Artvin Coruh University
Other Study IDs: EMG MS
Record Dates: First submitted 2025-11-15; First posted 2025-11-19 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; electromyography; urinary incontinence; pelvic floor; fatigue
MeSH Terms: conditions — Multiple Sclerosis; Urinary Incontinence; Fatigue

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Multiple Sclerosis (PwMS): Adults diagnosed with multiple sclerosis will be included in the study.

SUMMARY:
The study aimed to explore the link between urinary incontinence (UI) severity in patients with multiple sclerosis (PwMS), electromyography (EMG) findings, and other relevant factors.

DETAILED DESCRIPTION:
The study will consist of a cross-sectional observational analysis involving a cohort of 47 PwMS. The assessment will be employed various instruments, including the Expanded Disability Status Scale (EDSS), Neurogenic Bladder Symptom Score (NBSS), International Consultation on Incontinence Questionnaire Short Form (ICIQ-SF), Incontinence Impact Questionnaire (IIQ-7), International Physical Activity Questionnaire (IPAQ), Fatigue Severity Scale (FSS), EMG.

ELIGIBILITY:
Inclusion Criteria:

* having an MS diagnosis according to the 2017 revised McDonald criteria,
* experiencing symptoms of UI as defined by the International Continence Society (ICS),
* having an EDSS score below 6.5,
* PwMS with no communication issues.

Exclusion Criteria:

* PwMS who did not give consent to participate,
* those with medication changes in the past 6 months,
* pregnant PwMS,
* recent vaginal or caesarean deliveries within 6 months,
* pelvic organ prolapse,
* urinary tract infection,
* recent attack history in the past month.

Ages: 30 Years to 50 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — Only women with MS will be included.
Study Population: Women diagnosed with MS will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Expanded disability status scale (EDSS) | Single assessment at enrollment
  The Expanded disability status scale (EDSS) will be assessed disability and progression in PwMS, with scores from 0 (normal neurological exam) to 10 (death from MS). Higher scores indicate greater disability.
Neurogenic Bladder Symptom Score (NBSS) | Single assessment at enrollment
  Storage, voiding, and complication symptoms of neurogenic bladder will be assessed with the Neurogenic Bladder Symptom Score (NBSS), a 24-item questionnaire covering incontinence, storage and voiding, and outcomes.
International Consultation on Incontinence Questionnaire Short Form (ICIQ-SF) | Single assessment at enrollment
  The frequency and amount of leakage will be assessed using a six-item scale, and urinary incontinence will be categorised into four groups: mild (1-5), moderate (6-12), severe (13-18) and very severe.
Incontinence Impact Questionnaire (IIQ-7) | Single assessment at enrollment
  Urinary symptoms' impact on daily activities was assessed with the Incontinence Impact Questionnaire (IIQ-7). The 7-item Likert scale has a score range of 0-21, with higher scores reflecting an increased negative impact of incontinence on social functioning, quality of life, and physical activity.
Pelvic Floor Muscle Activity | Single assessment at enrollment
  An electromyography (EMG) device with surface electrodes will be used to assess pelvic floor muscle (PFM) activity. Patients received training beforehand, and measurements were taken noninvasively with two electrodes around the perineum and vagina and one on the inner thigh in women.
International Physical Activity Questionnaire (IPAQ) | Single assessment at enrollment
  The International Physical Activity Questionnaire (IPAQ) assesses the frequency and duration of vigorous, moderate, and walking-like activities over a week. The values are multiplied by factors of 8, 4, and 3.3 Metabolic Equivalent of Tasks, respectively, to help measure overall physical activity. The minimum score for the IPAQ is 0, while there is no theoretically determined maximum score. Higher scores are associated with the individual engaging in a higher level of physical activity.
Fatigue severity scale (FSS) | Single assessment at enrollment
  Fatigue severity scale (FSS) assesses fatigue severity in MS with nine items rated on a 7-point Likert scale. The mean score, adapted to Turkish society, indicates pathological fatigue if it is 4 or higher.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Yıldız Kızkın, Principal Investigator — Artvin Coruh University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zecca C, Riccitelli GC, Disanto G, Singh A, Digesu GA, Panicari L, Puccini F, Mattioli M, Tubaro A, Gobbi C. Urinary incontinence in multiple sclerosis: prevalence, severity and impact on patients' quality of life. Eur J Neurol. 2016 Jul;23(7):1228-34. doi: 10.1111/ene.13010. Epub 2016 Apr 27. PMID 27120000
- [Background] Tornic J, Panicker JN. The Management of Lower Urinary Tract Dysfunction in Multiple Sclerosis. Curr Neurol Neurosci Rep. 2018 Jun 28;18(8):54. doi: 10.1007/s11910-018-0857-z. PMID 29956001
- [Background] Afshari P, Abedi P, Majdinasab N, Tafakh S, Haghighizadeh M. Strengths of pelvic floor muscles in women with multiple sclerosis and its relationship with urinary incontinence and quality of life. Front Neurol. 2025 Jan 13;15:1514157. doi: 10.3389/fneur.2024.1514157. eCollection 2024. PMID 39871990